CLINICAL TRIAL: NCT05536609
Title: Cast Or ePineural Suture for Digital Nerve Injuries - a Randomised Controlled Study
Acronym: COPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Cecilia Mellstrand Navarro, MD PhD Ass prof, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COPS - RCT dig nerve injuries
Record Dates: First submitted 2022-08-23; First posted 2022-09-13 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Digital Nerve Injury
Keywords: digital nerve injury; digital nerve lesion; randomised controlled study; surgical nerve repair; non-operative treatment
MeSH Terms: interventions — Wound Healing; POLR1G protein, human

STUDY DESIGN:
Intervention Model Description: 1:1 randmoised controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epineural suture (Experimental): The injured digital nerve is exposed during a surgical intervention and sutured with 2 or three epineural sutures 8.0 or 9.0 synthetic monofilament non-resorbable suture. Postoperative treatment includes 3 weeks in a plaster cast followed by rehabilitation.
  Interventions: Procedure: Epineural suture
- Non-operative treatment (Active Comparator): The injured digital nerve is not surgically exposed. The skin is closed over the injury site and the finger is protected in a plaster cast for three weeks followed by rehabilitation.
  Interventions: Procedure: Non-operative treatment

INTERVENTIONS:
Procedure: Epineural suture — 2 or three sutures
  Other Names: surgical repair
  Arms: Epineural suture
Procedure: Non-operative treatment — The injured finger is protected in a plaster cast
  Other Names: cast
  Arms: Non-operative treatment

SUMMARY:
Nerve injury in the fingers is a common injury and affects people of all ages. The treatment usually offered to patients is surgery and various types of rehabilitation. There is a lack of knowledge and research on how these injuries should be treated in the best way and how well sensory function can be restored after an injury. In this research project, we will investigate results after treatment for digital nerve injuries by entailing a randomised controlled trial allocating patients with isolated digital nerve injuries to either surgical repair or non-operative treatment in a cast. Primary outcome is digital nerve function as measured by 2-points discrimination at 1 year after treatment. Secondary outcomes include finger mobility, dexterity, handfunction, occurence of pain and anxiety and time on sick leave.

DETAILED DESCRIPTION:
Patients over the age of 20 with an acute traumatic isolated digital nerve injury to any of the fingers and not in the thumb will be investigated for inclusion in the study. After informed written consent a sealed envelope randomisation will allocate patients to treatment with either surgical exposure and epineural suture or non-operative treatment in a cast. Due to the nature of treatment arms the allocation will not be blinded. Clinical follow-up and investigation of primary and secondary outcomes will be conducted at 3 weeks, 3 months, 6 months and 1 year after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs of isolated traumatic digital nerve injury in digits 2, 3, 4 or 5.
* Patient age => 20 years on day of injury.
* Injury location on volar aspect of finger.
* Acute sensory dysfunction in suspected digital nerve injury area.

Exclusion Criteria:

* Digital nerve injury ot the thumb
* Digital nerve injury in the palm of the hand (i e proximal to the finger base)
* Patient does not speak or read the Swedish language.
* Abusive drug or alcohol use
* Dementia.
* Injury mor than 7 days at dianosis AND/OR operative treatment cannot be offered within 10 days from injury.
* Neurologic disease.
* Ongoing infektion in the injured finger.
* concomittant tendoninjury or fracture in injured or adjacent finger.
* Injury mechanism is of blunt or crush charachter

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Static two points discrimination (S2PD) | one year after injury
  a static two points discrimination test performed by an occupational therapist of the injured finger

SECONDARY OUTCOMES:
Active range of motion | 3 and 6 months and 1 year
  Range of motion of the injured finger (sum of MCP + PIP + DIP joint motion measured in degrees)
Ratio between S2PD in injured finger and S2PD in uninjured contralateral finger | 3 and 6 months and 1 year
  Ratio between S2PD in injured finger and S2PD in uninjured contralateral finger
Semmes-Weinstein monofilament test | 3 and 6 months and 1 year
  Discriminatory sensory function as measured by Semmes-Weinstein monofilament test
Mini Sollerman test | 3 and 6 months and 1 year
  Hand function as measured by the Mini Sollerman test
Grip strength | 3 and 6 months and 1 year
  Grip strength of injured and non-injured hand as measured by Jamar dynamometer
Quick-DASH | 3 and 6 months and 1 year
  Patient Rated Outcome measure (PROM) for hand function as measured by the quick-DASH (Disability of the Arm, Shoulder and Hand). 11 items with 5-level Likert scales measures upper limb function. The scale ranges from 0 - 100 and 0 is the lowest possible disability.
HQ-8 | 3 and 6 months and 1 year
  Patient Rated Outcome measure (PROM) for hand function as measured by the HQ-8 (Eight item HAKIR questionnaire)
Neuropathic pain | 3 and 6 months and 1 year
  Occurrence of neuropathic pain as measured by Doleur Neuropathic 4 questions (DN4). 4 aspects of neuropathic pain are evaluated by 10 questions, with higher scores representing a worse state.
Anxiety and depression | at inclusion
  Psychologic wellbeing as measured by Hospital Anxiety and Depression scale (HAD) (PCS)
Pain catastrophising scale, (PCS) | at inclusion
  Pain catastrophising scale, (PCS) measures 13 items on a 5 points Likert scale. Higher scores represent high degree of pain catastrophising scale, (PCS).
Sick leave time | 1 year
  Days of absence from work
Wait for surgery | 3 weeks
  The number of days that have passed from the day of injury to the day of surgery are reported
Time in operating theatre | day of surgery
  Time in operating theatre is measured in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Mellstrand Navarro, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet Södersjukhuset, Department of clinical research and education, Stockholm, Stockholm County, Sweden